CLINICAL TRIAL: NCT07240753
Title: Clinical Characteristics and Prognostic Factors of Large Cell Neuroendocrine Carcinoma of the Cervix: A Multicenter, Bidirectional Cohort Study
Brief Title: A Chinese Cohort of Cervical Large Cell Neuroendocrine Carcinoma
Acronym: CN-CLCNEC
Status: Not yet recruiting | Type: Observational
Sponsor: Lili (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Cancer Research Institute of Zhongshan City (Other Government); The First Affiliated Hospital of Zhengzhou University (Other); Qilu Hospital of Shandong University (Other); Fujian Province Tumor Hospital (Other); Fujian Maternity and Child Health Hospital (Other); Zhejiang Cancer Hospital (Other); The Third Affiliated Hospital of Kunming Medical College. (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); Women's Hospital School Of Medicine Zhejiang University (Other); National Cancer Center/National Cancer Clinical Medical Research Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College (Unknown); Peking Union Medical College Hospital (Other); The Affiliated Tumor Hospital of Xinjiang Medical University (Unknown); The First Affiliated Hospital of Anhui Medical University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor-Investigator, Lili, Associate Chief Physician, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202506084
Record Dates: First submitted 2025-11-15; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-06

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Cervical Large Cell Neuroendocrine Carcinoma; Prognosis; High-Risk Factors; Treatment Options
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical Large Cell Neuroendocrine Carcinoma Cohort
  Interventions: Other: Postoperative pathological examination confirmed cervical large cell neuroendocrine carcinoma.

INTERVENTIONS:
Other: Postoperative pathological examination confirmed cervical large cell neuroendocrine carcinoma. — Postoperative pathological examination confirmed cervical large cell neuroendocrine carcinoma.

SUMMARY:
Cervical large cell neuroendocrine carcinoma (LCNEC) exhibits highly aggressive biological behavior, including strong invasiveness, a high propensity for metastasis, drug resistance, and poor prognosis, necessitating heightened clinical and pathological awareness. This study aims to summarize the clinical characteristics of LCNEC and analyze various prognostic factors to enhance understanding and vigilance toward this disease. Combined with precise pathological diagnosis, improving diagnostic accuracy is crucial for formulating treatment strategies and assessing patient prognosis.

DETAILED DESCRIPTION:
This study will collect the complete medical records of patients with cervical large cell neuroendocrine carcinoma registered in the participating tertiary hospitals, and will prospectively collect the medical records of patients diagnosed with cervical large cell carcinoma. The data to be collected includes:

* Patient demographics (age, place of origin, occupation, etc.)
* Medical history and test results prior to initial treatment:
* Present illness history
* Tumor marker levels
* Pelvic ultrasound
* Whole abdomen CT/MRI
* PET-CT
* Surgical treatment details (date of surgery, surgical approach)
* Pathological examination results
* Administration of neoadjuvant chemotherapy and/or radiotherapy
* Detailed records of all treatment courses and their efficacy (including chemotherapeutic agents, radiotherapy doses, number of cycles, etc.)
* Results from follow-up examinations and imaging studies
* Recurrence status and, if applicable, time to recurrence
* Survival status and, if applicable, date of death For the retrospective cohort, follow-up will be completed within one month after enrollment to document current survival status and recurrence. For the prospective cohort, annual follow-ups will be conducted to record current survival status and recurrence.

ELIGIBILITY:
Inclusion Criteria: The diagnosis of cervical large cell neuroendocrine carcinoma (LCNEC) was confirmed by histopathological examination, meeting both clinical and histological criteria. The tumor exhibited characteristic features, including large cells with abundant cytoplasm, vesicular nuclei with prominent nucleoli, and a high mitotic rate (>10 mitoses/10 HPFs). The growth patterns were predominantly insular, trabecular, or solid, often accompanied by peripheral palisading or rosette formation, along with focal tumor necrosis.

-

Exclusion Criteria: Mixed cervical LCNEC histology, cases with missing follow-up, or patients lost to contact.

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female patients diagnosed with cervical large cell neuroendocrine carcinoma by postoperative histopathological examination.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | One month post-enrollment completion and then annual follow-up
Disease Recurrence | One month post-enrollment completion and then annual follow-up

IPD SHARING:
Plan to Share IPD: Undecided
It involves highly confidential personal information.

REFERENCES:
- [Background] Takayanagi D, Hirose S, Kuno I, Asami Y, Murakami N, Matsuda M, Shimada Y, Sunami K, Komatsu M, Hamamoto R, Kato MK, Matsumoto K, Kohno T, Kato T, Shiraishi K, Yoshida H. Comparative Analysis of Genetic Alterations, HPV-Status, and PD-L1 Expression in Neuroendocrine Carcinomas of the Cervix. Cancers (Basel). 2021 Mar 10;13(6):1215. doi: 10.3390/cancers13061215. PMID 33802174
- [Background] Georgescu TA, Bohiltea RE, Munteanu O, Furtunescu F, Lisievici AC, Grigoriu C, Gherghiceanu F, Vladareanu EM, Berceanu C, Ducu I, Iordache AM. Emerging Therapeutic Concepts and Latest Diagnostic Advancements Regarding Neuroendocrine Tumors of the Gynecologic Tract. Medicina (Kaunas). 2021 Dec 7;57(12):1338. doi: 10.3390/medicina57121338. PMID 34946283
- [Background] Xu F, Yu Q, Wan D, Zhang Y. Cervical adenocarcinoma admixing with large cell neuroendocrine carcinoma: A rare case report. Asian J Surg. 2022 Dec;45(12):2932-2933. doi: 10.1016/j.asjsur.2022.06.109. Epub 2022 Jun 29. No abstract available. PMID 35778245
- [Background] Salvo G, Gonzalez Martin A, Gonzales NR, Frumovitz M. Updates and management algorithm for neuroendocrine tumors of the uterine cervix. Int J Gynecol Cancer. 2019 Jul;29(6):986-995. doi: 10.1136/ijgc-2019-000504. PMID 31263021
- [Background] Lee E, Ji YI. Large Cell Neuroendocrine Carcinoma of the Cervix with Sequential Metastasis to Different Sites: A Case Report. Case Rep Oncol. 2018 Oct 23;11(3):665-670. doi: 10.1159/000493912. eCollection 2018 Sep-Dec. PMID 30483095
- [Background] Caruso G, Sassu CM, Tomao F, Di Donato V, Perniola G, Fischetti M, Benedetti Panici P, Palaia I. The puzzle of gynecologic neuroendocrine carcinomas: State of the art and future directions. Crit Rev Oncol Hematol. 2021 Jun;162:103344. doi: 10.1016/j.critrevonc.2021.103344. Epub 2021 Apr 29. PMID 33933568